CLINICAL TRIAL: NCT04943900
Title: A Phase 1 Study of BMS-986416 Alone and in Combination With Nivolumab in Select Solid Tumors
Brief Title: A Study of BMS-986416 With and Without Nivolumab in Select Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA102-003
Record Dates: First submitted 2021-06-25; First posted 2021-06-29 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumors
Keywords: BMS-986416; Nivolumab; Opdivo; Non-small cell lung cancer (NSCLC); Urothelial carcinoma (UC); Squamous cell carcinoma of the head and neck (SCCHN); Hepatocellular carcinoma (HCC); Microsatellite-stable colorectal carcinoma (MSS CRC); Pancreatic ductal adenocarcinoma (PDAC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Transitional Cell; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Hepatocellular | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1A: Monotherapy (BMS-986416) (Experimental)
  Interventions: Drug: BMS-986416
- Part 1B: Combination Therapy (BMS-986416 + Nivolumab) (Experimental)
  Interventions: Drug: BMS-986416; Drug: Nivolumab

INTERVENTIONS:
Drug: BMS-986416 — Specified dose on specified days
Drug: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558; Opdivo
  Arms: Part 1B: Combination Therapy (BMS-986416 + Nivolumab)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, drug effects, drug levels and preliminary antitumor activity of BMS-986416 when administered alone and in combination with Nivolumab in participants with select advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically or cytologically confirmed locally advanced unresectable, metastatic, or recurrent select solid tumor
* Eligible tumor types Non-small cell lung cancer (NSCLC), Urothelial carcinoma (UC), Squamous cell carcinoma of the head and neck (SCCHN), Hepatocellular carcinoma (HCC), Microsatellite-stable colorectal carcinoma (MSS CRC), or Pancreatic ductal adenocarcinoma (PDAC)
* Resistant/refractory to or intolerant of existing standard therapies known to provide clinical benefit
* Measurable disease per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v 1.1)
* Disease amenable to serial biopsy

Exclusion Criteria:

* Uncontrolled or significant cardiovascular disease
* Known connective tissue disease such as Marfan, Ehlers-Danlos, or Loeys-Dietz syndrome
* Medical requirement for chronic anticoagulant or antiplatelet agents (except low-dose aspirin, which is permitted)

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 100 days after the last treatment of study intervention(s)
Incidence of Serious Adverse Events (SAEs) | Up to 100 days after the last treatment of study intervention(s)
Incidence of AEs meeting protocol-defined dose-limiting toxicity (DLT) criteria | Up to 100 days after the last treatment of study intervention(s)
Incidence of AEs leading to discontinuation | Up to 100 days after the last treatment of study intervention(s)
Incidence of AEs leading to death | Up to 100 days after the last treatment of study intervention(s)
Protocol-defined maximum tolerated dose (MTD) or maximum administered dose (MAAD) | Up to 100 days after the last treatment of study intervention(s)

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) of BMS-986416 | Up to 100 days after the last treatment of study intervention(s)
Time of maximum observed serum concentration (Tmax) of BMS-986416 | Up to 100 days after the last treatment of study intervention(s)
Trough observed serum concentration (Ctrough) of BMS-986416 | Up to 100 days after the last treatment of study intervention(s)
Overall Response Rate (ORR) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) per Investigator assessment | Up to 2 years
Duration of Response (DOR) using RECIST 1.1 per Investigator assessment | Up to 2 years
Incidence of clinically significant changes in ECG parameters: QTcF | Up to 100 days after the last treatment of study intervention(s)
  QTcF = Corrected QT interval using the Fridericia formula. QT interval is the time from the start of the Q wave to the end of the T wave

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (19):
- United States (6):
  - Local Institution - 0006, Atlanta, Georgia
  - Local Institution - 0005, Baltimore, Maryland
  - Local Institution - 0002, Hackensack, New Jersey
  - Local Institution - 0013, Cleveland, Ohio
  - Local Institution - 0003, Pittsburgh, Pennsylvania
  - Local Institution - 0004, Houston, Texas
- Argentina (3):
  - Local Institution - 0021, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0027, ABB, Buenos Aires F.D.
  - Local Institution - 0022, CABA, Buenos Aires F.D.
- Belgium (2):
  - Local Institution - 0043, Edegem, Antwerpen
  - Local Institution - 0016, Ghent, Oost-Vlaanderen
- Canada (3):
  - Local Institution - 0009, Edmonton, Alberta
  - Local Institution - 0008, Toronto, Ontario
  - Local Institution - 0001, Montreal, Quebec
- Chile (3):
  - Local Institution - 0025, Santiago, Santiago Metropolitan
  - Local Institution - 0026, Santiago, Santiago Metropolitan
  - Local Institution - 0024, Santiago, Santiago Metropolitan
- Local Institution - 0010, Chuo-ku, Tokyo, Japan
- Local Institution - 0020, Maastricht, Limburg, Netherlands

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com